CLINICAL TRIAL: NCT05377060
Title: Disclosing Dementia Risk Based on Plasma Phosphorylated Tau
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Corey Bolton, Postdoctoral Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 220449
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma p-tau Disclosure (Experimental): To receive risk estimate based on plasma p-tau results in addition to age, sex, and cognitive screening score.
  Interventions: Behavioral: Plasma p-tau risk disclosure
- Standard Disclosure (Active Comparator): To receive risk estimate based on age, sex, and cognitive screening score.
  Interventions: Behavioral: Standard risk disclosure

INTERVENTIONS:
Behavioral: Plasma p-tau risk disclosure — Participants will receive an estimated risk for converting to dementia in the next four years based on age, sex, MMSE score, and plasma p-tau results.
  Arms: Plasma p-tau Disclosure
Behavioral: Standard risk disclosure — Participants will receive an estimated risk for converting to dementia in the next four years based on age, sex, and MMSE score.
  Arms: Standard Disclosure

SUMMARY:
Novel blood-based biomarkers of Alzheimer's disease (AD), such as plasma levels of tau phosphorylated at threonine 181 (p-tau181), have shown great promise in detecting early AD pathology. While current studies point to this biomarker as having great clinical utility, one necessary step before clinical implementation is developing safe and effective methods for disclosure of results. Past risk disclosure studies have shown that disclosing risk for AD based on genetics or amyloid status is safe, but these studies have largely focused on cognitively unimpaired individuals. This study seeks to develop comprehensible educational materials to aid risk disclosure and examine the effect of risk disclosure based on plasma p-tau181 results in a group of participants with mild cognitive impairment (MCI) at imminent risk of converting to dementia. First, educational materials will be developed in collaboration with health communication experts and then refined in focus groups made up of individuals with MCI. Educational materials will be analyzed on several key reading and comprehensibility metrics and will include personalized risk estimate based on a well-accepted risk algorithm (Cullen, et al., 2021). Next, these educational materials will be utilized to disclose risk in a randomized controlled trial with an active control arm receiving disclosure based on age, sex, and cognitive status (based on Mini-Mental State Examination), meant to mimic common methods of clinical diagnostic and prognostic decision making, and an intervention arm receiving disclosure based on the above factors plus plasma p-tau181 results. Outcomes will include measures of comprehension and psychological well-being (anxiety, depression, hopelessness, and distress) and will be assessed immediately after risk disclosure and again at six-month follow-up. It is hypothesized that risk disclosure based on plasma p-tau181 is not more psychologically harmful or less comprehensible than disclosure based on demographic factors and MMSE. This pilot study will provide a necessary step towards moving plasma p-tau biomarkers towards safe clinical implementation and will develop educational materials that can be utilized in future studies and clinical practice.

DETAILED DESCRIPTION:
Novel blood-based biomarkers of Alzheimer's disease (AD), such as plasma levels of tau phosphorylated at threonine 181 (p-tau181), have shown great promise in sensitively and specifically detecting early AD pathology. Plasma p-tau181 has the potential to dramatically reduce the financial strain and patient care burden associated with identifying patients at increased risk of AD-dementia, as well as improve screening for enrollment in clinical trials which require the presence of AD-pathological changes. While current studies point to this biomarker as having great clinical utility, one necessary step before clinical implementation is developing safe and effective methods for disclosure of results. Past risk disclosure studies have shown that disclosing risk for AD based on genetics or amyloid status is safe, but these studies have largely focused on cognitively unimpaired individuals. This study seeks to develop comprehensible educational materials to aid risk disclosure and examine the effect of risk disclosure based on plasma p-tau181 results in a group of participants with mild cognitive impairment (MCI) at imminent risk of converting to dementia. First, educational materials will be developed in collaboration with health communication experts and then refined in focus groups made up of individuals with MCI. Educational materials will be analyzed on several key reading and comprehensibility metrics and will include personalized risk estimate based on a well-accepted risk algorithm (Cullen, et al., 2021). Next, these educational materials will be utilized to disclose risk in a randomized controlled trial with an active control arm receiving disclosure based on age, sex, and cognitive status (based on Mini-Mental State Examination), meant to mimic common methods of clinical diagnostic and prognostic decision making, and an intervention arm receiving disclosure based on the above factors plus plasma p-tau181 results. Outcomes will include measures of comprehension and psychological well-being (anxiety, depression, hopelessness, and distress) and will be assessed immediately after risk disclosure and again at six-month follow-up. It is hypothesized that risk disclosure based on plasma p-tau181 is not more psychologically harmful or less comprehensible than disclosure based on demographic factors and MMSE. This pilot study will provide a necessary step towards moving plasma p-tau biomarkers towards safe clinical implementation and will develop educational materials that can be utilized in future studies and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants recruited will include 62 adults aged 60 and older.
2. Consensus diagnosis of amnestic MCI by Vanderbilt Alzheimer's Disease Research Center (VADRC) clinician panel.
3. Availability of a reliable study partner (reliable is defined as someone who interacts significantly with the participant and is available to participate in study visits in person).
4. English language fluency.

Exclusion Criteria:

1. Individuals who lack decisional capacity to provide informed consent at baseline will not be enrolled in the study.
2. History of major psychiatric illness (e.g., schizophrenia, bipolar), neurological illness (e.g., epilepsy, multiple sclerosis, Parkinson's disease), or head injury with significant loss of consciousness.
3. Presence of acute psychological distress (i.e., Geriatric Depression Scale >10 at screening).
4. Participation in other risk disclosure protocols.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale | Immediately following disclosure
  Questionnaire assessing depression
Geriatric Depression Scale - 6-month follow-up | Immediately following disclosure and at 6-month follow-up
  Questionnaire assessing depression
Geriatric Anxiety Scale | Immediately following disclosure
  Questionnaire assessing anxiety
Geriatric Anxiety Scale - 6-month follow-up | At 6-month follow-up
  Questionnaire assessing anxiety
Beck Hopelessness Scale | Immediately following disclosure
  Questionnaire assessing hopelessness
Beck Hopelessness Scale - 6-month follow-up | At 6-month follow-up
  Questionnaire assessing hopelessness
Impact of Events Scale | At 6-month follow-up
  Questionnaire assessing event-related distress
Immediate Comprehension | Immediately following disclosure
  Semi-structured interview to assess comprehension of disclosure information
Long-term Comprehension | At 6-month follow-up
  Semi-structured interview to assess comprehension of disclosure information

CONTACTS AND LOCATIONS:
Overall Officials: Corey J Bolton, PsyD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No